CLINICAL TRIAL: NCT07377266
Title: The Impact of Changing to a New Child- and Family-centered Outpatient Diabetes Clinic Focusing on Early Involvement of the Child With Diabetes, Training in Calmness Around Diabetes Management, Healthy Lifestyle, and Creating Peer-to-peer Networks
Acronym: StenoChild
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Nanna Lind, Post doctoral researcher, PhD, RN, Steno Diabetes Center Copenhagen
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H-25016032; p-2024-17600 (Other: Danish Data Protection Agency)
Record Dates: First submitted 2026-01-13; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Diabetes; Quality of Life; Children
Keywords: Diabetes; Children; Quality of Life; peer support; Play; Calmness; Group-based education
MeSH Terms: conditions — Diabetes Mellitus | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- StenoChild intervention (Experimental): See below, Families are randomized pragmatically based on their assigned HCP. Approximately 50% will attend a new clinic offering group-based, family-centered care (90-100 families); the rest receive standard care, with the intervention offered later in a waitlist design.
  Interventions: Behavioral: Group consultations and peer-to-peer learning
- Standard Care (Placebo Comparator): Families are randomized pragmatically based on their assigned HCP. Approximately 50% will attend a new clinic offering group-based, family-centered care (90-100 families); the rest receive standard care, with the intervention offered later in a waitlist design.
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Behavioral: Group consultations and peer-to-peer learning — The intervention introduces strategies to promote structured meals, calmness, and balanced diabetes self-management using play and storytelling learning strategies.
  Families participate in interactive modules in small groups (~6-8 families), covering topics like "Meal Calmness" and "Calm Mind" four times during a year (every third month). Parents learn practical techniques to reduce conflict and improve dialogue around diabetes management. Children under 7 receive play-based sessions; those 7 and older receive story-based sessions.
  Clinical data as well as questionnaires will be collected at each session.
  Arms: StenoChild intervention
Other: Standard Care (in control arm) — The control group receives standard care, with the intervention offered later in a waitlist design.
  Clinical data as well as questionnaires will be collected at baseline and again after one year.
  Arms: Standard Care

SUMMARY:
The goal of StenoChild is to strengthen the treatment of children under 10 years old with diabetes through a multi-component approach. This includes play-based methods, a focus on nutrition and mental health, and peer-to-peer programs that facilitate parental support and learning. The project has both a clinical and organizational dimension, as it aims to improve diabetes care and change practices and task organization at Steno Diabetes Center Copenhagen, SDCC.

DETAILED DESCRIPTION:
The investigators encourage families to engage in eating, exercising, playing, and storytelling together, leveraging children's natural inclination to learn through play. This approach allows healthcare providers (HCPs) and parents to gain insights into the child's perspective, improving communication.

The hypotheses are i) improved calmness during diabetes-related tasks with potential painful procedures such as shift of insulin infusions set and sensor will ease diabetes management and reduce parental distress; ii) improved structure and calmness around meals will ease diabetes management, reflected in interaction with insulin pumps; iii) the group and play-based approach will lead to healthier lifestyle changes compared to usual care.

ELIGIBILITY:
Inclusion of children and their families

Inclusion Criteria:

* Age 3-10 years
* Followed at Steno Diabetes Center Copenhagen

Exclusion Criteria:

* Severe psychiatric disease
* Language barriers (Children not speaking Danish, Parents not speaking Danish or English)

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Parental diabetes-related quality of life (T1DAL) | From baseline to study end after one year
  Change in Parental diabetes-related quality of life, measured by the questionnaire T1DAL in Danish. An increase in score indicates an improvement in parental diabetes-related quality of life.
Children's perception of clinical visits (MyHospitalVoice) | From baseline to study end after one year
  Change in Children's perception of clinical visits, measured by the questionnaire MyHospitalVoice in Danish. An increase in score indicates an improvement in perception of clinical visits-

SECONDARY OUTCOMES:
Change in glycemic outcomes by CGM-derived metrics | From baseline to study end after one year
  Time in range (glucose levels 3.9-10 mmol/l), time above range (>10 mmol/l), time below range (<3.9 mmol/l), in percentages of time, measured over the last 14 days.
Change in glycemic outcomes measured by HbA1c | From baseline to study end after one year
  Hba1c in mmol/mol
Change in total daily dose of insulin per kg | From baseline to study end after one year
  Measured as a mean value during the last 14 days
Change in the number of boluses registered per day | From baseline to study end after one year
  registered by the insulin pump, measured as a mean value during the last 14 days
Change in timing of boluses | From baseline to study end after one year
  Missed or late boluses registered by the insulin pump. Measured as a mean value during the last 14 days
Change in carbohydrates/kg entered per day | From baseline to study end after one year
  Registered by the insulin pump. Measured as a mean value during the last 14 days
Change in infusion set wear-time | From baseline to study end after one year
  Registered by the insulin pump. Measured as a mean value during the last 14 days
Change in time in automated insulin delivery mode (AID) on the insulin pump system. | From baseline to study end after one year
  Registered by the insulin pump, in percentages of time during the last 14 days.
Change in conflicts and problems with procedures | From baseline to study end after one year
  Change in conflicts around meals; FLACC (pain and fear scores and conflicts around painful procedures related to diabetes management)
Change in parental fear of hypoglycemia | From baseline to study end after one year
  Change in parental fear of hypoglycemia measured by questionnaire
Change in BMI z-scores | From baseline to study end after one year
  Age, sex, weight, and height will be used to report BMI z-scores for children by using WHO definitions for children in the age; 0-5 and 5-10 years.
Participation in planned modules | From baseline to study end after one year
  Participation pr. year pr. family out of the four held modules.

CONTACTS AND LOCATIONS:
Overall Officials: Jannet Svensson, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No